CLINICAL TRIAL: NCT03216668
Title: A Randomized, Active-Control, Open Label, Phase IIIb Study to Evaluate the Safety and Efficacy of TONKA Compared With Silymarin (Legalon) for Lowering Hepatic Enzymes in Liver Function Disorder Patients With Moderate to High Elevated Liver
Brief Title: TONKA Versus Legalon for Lowering Hepatic Enzymes in Liver Function Disorder Patients.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nhat Nhat Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TONKA-V3
Record Dates: First submitted 2017-07-09; First posted 2017-07-13 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Liver Function Failure
MeSH Terms: conditions — Hepatic Insufficiency | interventions — Silymarin

STUDY DESIGN:
Intervention Model Description: Block randomization
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TONKA (Experimental): Administered orally twice a day, 2 tablets each time, for 6 weeks
  Interventions: Drug: TONKA
- LEGALON (Active Comparator): Administered orally three times a day, two tablets each time, for 6 weeks
  Interventions: Drug: LEGALON

INTERVENTIONS:
Drug: TONKA — Administered orally twice a day, 2 tablets each time, for 6 weeks.
  Arms: TONKA
Drug: LEGALON — Administered orally three times a day, two tablets each time, for 6 weeks
  Arms: LEGALON

SUMMARY:
The purpose of this study is to evaluate the efficacy TONKA on the reduction of ALT and AST in moderate to severe liver enzyme elevated patients; compared with Silymarin (Legalon) after 6 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female more than 18 year old.
* Diagnosed as Alcoholic Liver Disease (ALD), or Non Alcoholic Fatty Liver Disease (NAFLD), or Liver Function Disorders due to Drugs or Chemicals.
* ALT at baseline is in between 150 U/L to 400 U/L
* Sign the informed consent form

Exclusion Criteria:

* Hepatitis B or C.
* Pregnant or Lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with ALT reduced to less than or equal to 60 U/L after 6 weeks of treatment, compared between Tonka and Silymarin (Legalon) | 6 weeks

SECONDARY OUTCOMES:
The percentage of patients with ALT reduced to less than or equal to 40 U/L after 3 weeks of treatment, compared between Tonka and Silymarin (Legalon) | 3 weeks
The percentage of patients with ALT reduced to less than or equal to 40 U/L after 6 weeks of treatment, compared between Tonka and Silymarin (Legalon) | 6 weeks
The percentage of patients with AST reduced to less than or equal to 40 U/L after 3 weeks of treatment, compared between Tonka and Silymarin (Legalon) | 3 weeks
The percentage of patients with AST reduced to less than or equal to 40 U/L after 6 weeks of treatment, compared between Tonka and Silymarin (Legalon) | 6 weeks
The percentage of patients with GGT reduced to less than or equal to 40 U/L after 3 weeks of treatment, compared between Tonka and Silymarin (Legalon) | 3 weeks
The percentage of patients with GGT reduced to less than or equal to 40 U/L after 6 weeks of treatment, compared between Tonka and Silymarin (Legalon) | 6 weeks
The percentage of patients with Total Bilirubin reduced to less than or equal to the upper normal limit (UNL) after 3 weeks of treatment, compared between Tonka and Silymarin (Legalon) | 3 weeks
The percentage of patients with Total Bilirubin reduced to less than or equal to the upper normal limit (UNL) after 6 weeks of treatment, compared between Tonka and Silymarin (Legalon) | 6 weeks
The percentage of patients with ALT reduced to less than or equal to 80 U/L after 3 weeks of treatment, compared between Tonka and Silymarin (Legalon) | 3 weeks
The percentage of patients with ALT reduced to less than or equal to 80 U/L after 6 weeks of treatment, compared between Tonka and Silymarin (Legalon) | 6 weeks
The percentage of patients with AST reduced to less than or equal to 80 U/L after 3 weeks of treatment, compared between Tonka and Silymarin (Legalon) | 3 weeks
The percentage of patients with AST reduced to less than or equal to 80 U/L after 6 weeks of treatment, compared between Tonka and Silymarin (Legalon) | 6 weeks
The percentage of patients with GGT reduced to less than or equal to 80 U/L after 3 weeks of treatment, compared between Tonka and Silymarin (Legalon) | 3 weeks
The percentage of patients with GGT reduced to less than or equal to 80 U/L after 6 weeks of treatment, compared between Tonka and Silymarin (Legalon) | 6 weeks
The percentage of patients with Total Bilirubin reduced to less than or equal to the 2 times of the upper normal limit (2xUNL) after 3 weeks of treatment, compared between Tonka and Silymarin (Legalon) | 3 weeks
The percentage of patients with Total Bilirubin reduced to less than or equal to the 2 times of the upper normal limit (2xUNL) after 6 weeks of treatment, compared between Tonka and Silymarin (Legalon) | 6 weeks
The absolute change from Baseline to 3 weeks in ALT, compared between Tonka and Silymarin (Legalon) | 3 weeks
The absolute change from Baseline to 6 weeks in ALT, compared between Tonka and Silymarin (Legalon) | 6 weeks
The absolute change from Baseline to 3 weeks in AST, compared between Tonka and Silymarin (Legalon) | 3 weeks
The absolute change from Baseline to 6 weeks in AST, compared between Tonka and Silymarin (Legalon) | 6 weeks
The absolute change from Baseline to 3 weeks in GGT, compared between Tonka and Silymarin (Legalon) | 3 weeks
The absolute change from Baseline to 6 weeks in GGT, compared between Tonka and Silymarin (Legalon) | 6 weeks
The absolute change from Baseline to 3 weeks in Total Bilirubin, compared between Tonka and Silymarin (Legalon) | 3 weeks
The absolute change from Baseline to 6 weeks in Total Bilirubin, compared between Tonka and Silymarin (Legalon) | 6 weeks
The number of participants with other clinically significant laboratory parameters at week 6, compared between Tonka and Silymarin (Legalon). | 6 weeks
The number of participants with clinically significant vital sign parameters at week 6, compared between Tonka and Silymarin (Legalon). | 6 weeks

OTHER OUTCOMES:
The absolute change after treatment discontinuation from week 6 to week 10 in ALT , compared between Tonka and Silymarin (Legalon) | week 6, week 10
The absolute change after treatment discontinuation from week 6 to week 10 in AST , compared between Tonka and Silymarin (Legalon) | week 6, week 10
The absolute change after treatment discontinuation from week 6 to week 10 in GGT , compared between Tonka and Silymarin (Legalon) | week 6, week 10
The absolute change after treatment discontinuation from week 6 to week 10 in Total Bilirubin, compared between Tonka and Silymarin (Legalon) | week 6, week 10

CONTACTS AND LOCATIONS:
Locations (1):
- Hue Central General Hospital, Huế, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided